CLINICAL TRIAL: NCT04454073
Title: Investigation of Factors Associated With Preserved Cognitive Function in Bipolar Disorder
Status: Active, not recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 67144
Record Dates: First submitted 2020-06-08; First posted 2020-07-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Disorder
Keywords: Cognition; Cross-sectional Studies
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bipolar patients: In euthymic state or with mild to moderate symptoms

SUMMARY:
Bipolar disorder (BD) ïs the fourth leading cause of disability worldwide among young people. Differences in demographic and clinical characteristics between patients do not influence educational achievement and receipt of disability pension, indicating that there are other factors such as neurocognitive function that are of importance for maintaining occupational and social function. Research has shown that at the group level, cognitive deficits are present in euthymic BD patients, while approximately 30%-50% of BD patients is not different from healthy controls when it comes to cognitive function. There is however little knowledge of risk and resilience factors for cognitive impairment in BD. Factors likely to contribute to cognitive and functional outcomes in BD, such as sleep, obesity, biological rhythms, comorbid medical and psychiatric conditions are also understudied. While it has been customary to focus research on factors related to the negative illness trajectories, the overarching aim of the current project is to explore factors associated with favourable outcomes. This shift in research focus is essential to elucidate factors related to more preserved function since this represents a clear gap in knowledge today.

DETAILED DESCRIPTION:
This is an observational and prospective study aimed at identifying risk and resilience factors for cognitive impairment in BD. The investigators will enrol 85 participants with bipolar disorder. The assessment period is from one up to two weeks. At inclusion, the investigators will examine other psychiatric conditions, known somatic diseases and symptom levels of depression and hypo-/mania. Insomnia severity and risk factors for metabolic syndrome will also be assessed. Secondly, the investigators will examine sleep and Activity extensively with both subjective and objective measures for one to two weeks. Third, a newly developed web-based neuropsychological test protocol will be used shortly after assessment of sleep and activity to test cognitive function. Fourth, alcohol use, substance use and biological rhythms will be assessed. Lastly, the investigators will retest cognitive function and symptom levels up to five years after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged >=18 years who score <= 16 on the MADRS or <= 8 on the YMRS.
* Willing and able to give online informed consent.

Exclusion Criteria:

* Symptom level above inclusion criteria will be put on a waiting list, and if informed consent is given, will be included when symptom level is reduced.
* No Norwegian fluency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bipolar patients diagnosed with Bipolar disorder I or II, in euthymic state or with mild to moderate symptoms at time of assessment.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of cognitive function in bipolar patients | On day 7 after inclusion
  Memoro is a self-administered web-based neuropsychological test platform. All tests include both written and auditory instructions. The Memoro will be used to assess objective cognitive function. It contains measures of learning, storing, recalling and recognizing visual and verbal information, pattern separation, and verbal memory span, verbal working memory, processing speed, reaction time and cognitive control. Time frame: After examination of sleep and activity for a period of up to two weeks. Results from the test will be converted to z-scores.
Assessing change of cognitive function in bipolar patients | Up to 5 years after inclusion
  Memoro is a self-administered web-based neuropsychological test platform. All tests include both written and auditory instructions. It contains measures of learning, storing, recalling and recognizing visual and verbal information, pattern separation, and verbal memory span, verbal working memory, processing speed, reaction time and cognitive control. The Memoro will be used to assess stability or change in objective cognitive function.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale (MADRS) | Day 1
  MADRS will be used to assess depressive symptoms. Range is 0-60. Higher score indicate more severe depressive symptoms.
Young Mania Rating Scale (YMRS) | Day 1
  YMRS will be used to assess hypo-/manic symptoms. Range is 0 to 60. Higher score indicate more severe manic symptoms.
Insomnia Severity Index (ISI) | Day 1
  A self-reported questionnaire of insomnia severity. Range is 08-28. Higher values represent higher levels of insomnia symptom severity.
Medication use | Day 1
  Daily doses and classes of medications (e.g. antipsychotics, mood stabilizers, benzodiazepines, etc.) prescribed per individual by the time of inclusion will be recorded.
Actigraph | 1 week
  Actigraph is a small device usually worn on the wrist that records the activity level of the body by sensing physical movement. The actigraph will be used to objectively assess sleep variables and daytime activity parameters.
Sleep diary | 1 week
  A self-reported record of the participants' sleeping and waking times.
Oximetry | 1 day (1 night during period of sleep assessment)
  Oximetry is a measurement of the blood's oxygen saturation. It will be used to assess any indication of sleep apnea for one night during the period of sleep assessment
The Functioning Assessment Short Test (FAST) | 7 days after inclusion
  FAST will be used to assess functional outcomes. Range is 0-72. Higher values indicate greater disability
Cognitive complaints in Bipolar disorder Rating Assessment (COBRA) | 7 days after inclusion
  COBRA is an assessment of subjective cognitive dysfunction. Range is 0-48 and higher scores indicate more cognitive complaints.
The Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN) | 7 days after inclusion
  BRIAN is an assessment of circadian rhythms disturbance. Range is 1 to 72 and higher score indicate more severe disturbance of circadian rhythms.
Alcohol use disorders identification test (AUDIT) | 7 days after inclusion
  AUDIT is an assessment of the frequency and quantity of alcohol consumption where higher scores indicate higher levels of use.
Drug use disorders identification test (DUDIT) | 7 days after inclusion
  DUDIT is an assessment of the frequency and quantity of drug consumption where higher scores indicate higher levels of use.
Number of participants With Metabolic syndrome | 7 days after inclusion
  The World Health Organisation criteria for the metabolic syndrome will be used in the dichotomisation of the metabolic factors: Systolic blood pressure will be dichotomised as ≤ 140 mmHg or >140 mmHg and diastolic blood pressure as ≤ 90 mmHg or > 90 mmHg. Triglycerides will be classified as < 1.7 mmol/l or ≥ 1.7mmol/l. HDL cholesterol will be categorised as ≥ 1 mmol/l or <1 mmol/l for women and ≥ 0.90 mmol/l or <0.90 mmol/l for men. Fasting glucose will be defined as elevated when the plasma glucose levels is ≥7.0 mmol/l and two dichotomous groups will be created; < 7.0 mmol/l or ≥ 7.0 mmol/l. Waist circumference will be measured at the level of the umbilicus, and the hip girth will be measured at the level of maximal protrusion of the gluteal muscles. Waist-to-hip ratio will be dichotomised as ≤ 0.85 or > 0.85 for women and ≤ 0.90 or > 0.90 for men. The waist circumference will be categorised as ≤ 88 cm or > 0.88 for women and ≤ 102 cm or >102 cm for men.
Numbers of participants With disturbances of Thyroid function | 7 days after inclusion
  Normal thyroid function is considered thyroid stimulating hormone (TSH) levels in the range from 0.24 to 3.78 mIU/l and T4 levels in the range of 13.5 to 21.2 pmol/l.
  Latent and subclinical biochemical hypothyroidism; with an elevation of TSH with T4 in the normal range.
  Overt biochemical hypothyroidism: elevated TSH and a decrease of T4 levels. Biochemical hyperthyroidism and latent biochemical hyperthyroidism: TSH levels below the normal range with and without elevated T4.
Diagnostic evaluation With Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-5) | Day 1
  This measure will be used to determine if participants meet the diagnostic criteria for Bipolar Disorder. This is a yes/no diagnostic tool and our data indicate percentage who meet criteria for bipolar type I or type II.

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Vestvik, Study Director — St Olavs Hospital, Division of Mental Health Care; Anne Engum, phd, Principal Investigator — St Olavs Hospital, Division of Mental Health Care; Knut Langsrud, Study Director — St Olavs Hospital, Division of Mental Health Care
Locations (1):
- Bipolar and sleep outpatient clinic, Department of Østmarka, Division of Mental Health Care, Trondheim, Norway

REFERENCES:
- [Derived] Svee K, Morken G, Hansen TI, Engum A. Internet-Based Cognitive Assessments During Remission in Bipolar Disorder: Subjective Cognitive Function and Clinical Severity. Acta Psychiatr Scand. 2025 Aug 31. doi: 10.1111/acps.70031. Online ahead of print. PMID 40887748